CLINICAL TRIAL: NCT05758896
Title: Effect on Contrast Induced Acute Kidney Injury of APX-115 in Subjects Undergoing Percutaneous Coronary Intervention A Randomized, Double-blind, Parallel Group, Multicenter, Multi-national Trial
Brief Title: Study of APX-115 in Contrast Induced Acute Kidney Injury in Subjects Undergoing PCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aptabio Therapeutics, Inc. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A01-115-04
Record Dates: First submitted 2022-05-27; First posted 2023-03-08 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Contrast Induced Acute Kidney Injury
Keywords: Isuzinaxib; APX-115; Contrast media; ROS; Acute Kidney Injury; Percutaneous Coronary Intervention
MeSH Terms: conditions — Acute Kidney Injury | interventions — isuzinaxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Isuzinaxib (APX-115) (Experimental): 4 x Isuzinaxib 88 mg calculated as free base (4 x 100mg APX-115(Isuzinaxib hydrocloride) capsules as salt form) administered QD, orally, for 5 consecutive days
  Interventions: Drug: Isuzinaxib (APX-115)
- Placebo (Placebo Comparator): 4 x Placebo capsules administered QD, orally, for 5 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isuzinaxib (APX-115) — Treatment allocation in 1:1 ratio to Isuzinaxib or Placebo
  Other Names: Isuzinaxib Hydrochloride
  Arms: Isuzinaxib (APX-115)
Drug: Placebo — Treatment allocation in 1:1 ratio to Isuzinaxib or Placebo
  Arms: Placebo

SUMMARY:
This phase 2 study is to assess the safety and efficacy of APX-115 active doses in Contrast Induced Acute Kidney Disease compared to placebo following multiple oral dosing in patients with undergoing percutaneous coronary intervention. It is anticipated that approximately 280 patients will be randomized into the study in a 1:1 ratio to 400 mg APX-115 (Isuzinaxib hydrochloride) or placebo arm.

DETAILED DESCRIPTION:
Patients with chronic kidney disease undergoing percutaneous coronary intervention deserve careful consideration of various clinical options to minimize the risk of contrast-induced acute kidney injury and to optimize clinical outcomes. Contrast-induced acute kidney injury (CI-AKI) is a leading cause of a hospital-acquired renal failure and has been reported to affect both the mortality and morbidity of patients receiving contrast media. Contrast-induced acute kidney injury is the third leading cause of hospital-acquired acute kidney injury and has been recognized as a serious complication of percutaneous coronary intervention (PCI), which may be associated with increased morbidity and mortality.

APX-115 is a potent small molecule inhibitor of NADPH-oxidase (NOX) isozymes developed by AptaBio Therapeutics, Inc. In-vivo study results suggest that multiple NOX isoforms may contribute to renal injury in CI-AKI model, and pan-NOX inhibition may be a new therapeutic approach for prevention of CI-AKI.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent.
2. Male or female, of any race or ethnicity, 18 years of age or older, inclusive, on the day of informed consent. Racial and ethnic minorities should be included in the study population to the greatest extent possible.
3. Diagnosed with coronary artery disease.
4. Planned to undergo coronary angiography within 4 weeks of being consented.
5. Risk of CKD evidenced by 30 mL/min/1.73m2 ≤ eGFR (Glomerular filtration rate) < 90 mL/min/1.73 m2 confirmed by local or central laboratory.
6. Women of childbearing potential or males willing and able to use at least one protocol-specified method of contraception for the duration of their enrolment.
7. Subject is aware of the investigational nature of this study and willing to comply with protocol treatments, blood tests, and other evaluations listed in the ICF.

Exclusion Criteria:

1. Females who are pregnant or who are planning to become pregnant before the end of planned enrolment or who are breastfeeding.
2. Subjects who are not expected to go through PCI at the discretion of investigator or cardiologist
3. Subjects who have a history of hypersensitivity to contrast media or who cannot be administered contrast media according to investigator's discretion
4. Acute myocardial infarction within 1 month prior to Screening
5. ESRD confirmed by eGFR < 15 mL/min/1.73 m2 at Screening.
6. Clinically significant heart disease as determined by the Investigator within 2 months prior to Screening including but not limited to any of following; cardiogenic shock, treatment requiring intra-aortic balloon pump (IABP) support, treatment with extra corporeal membrane oxygenation (ECMO), or NYHA class IV heart failure.
7. Uncontrolled treated/untreated hypertension (defined as systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg, mean of measured 2 times at Screening will be permitted).
8. Known or suspected hypersensitivity to any component of the APX-115 formulation.
9. History of acute kidney injury or renal dialysis within 1 month prior to Screening and/or plan to undergo a renal dialysis during enrolment.
10. Clinically apparent liver disease as determined by the Investigator (e.g., jaundice, cholestasis, hepatic synthetic impairment, or active hepatitis) or moderate or severe hepatic impairment as determined by Child-Pugh score (Class B or C) at Screening.
11. Impaired liver function, defined as alanine aminotransferase (ALT) ≥ 2.5 times UNL or Total bilirubin >1.5 × ULN, unless the subject has known Gilbert's syndrome.
12. Any sign or symptom of acute or chronic infection at Screening.
13. Receipt of any investigational drug within 4 weeks prior to Screening.
14. Confirmed or suspected abuse of alcohol or controlled substances within 1 year prior to Screening.
15. Clinically significant hematology abnormalities; hemoglobin <9 g/dL for females or <11 g/dL for males, absolute neutrophil count <1500/mm3, platelet count <100 × 109/L) at Screening. If any parameter is below the specified threshold, one hematology retest analyzed at the central or local laboratory within a week prior to randomization is permitted with the result of the last sample being conclusive.
16. Any other clinically significant medical condition or laboratory abnormality as determined by the Investigator that might jeopardize the safety of the subject, impair subject compliance, or impede safety/efficacy observations during enrolment.
17. Mental incapacity, unwillingness, or language barrier precluding adequate understanding or cooperation with protocol requirements
18. Use of CYP1A2, CYP2B6 and CYP3A4 substrates or UGT inhibitors and inducers or OAT3 substrates prior to enrollment or concurrently. It will be only accepted to be eligible to screening if the subjects' concomitant medications will be reviewed and approved by the medical monitor and/or sponsor prior to the initial study dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety endpoints: adverse event | Day -2 to day 84
  Number of adverse events
Safety endpoints: vital sign | Day 0 to day 84
  Number of subjects with abnormal Vital Signs
Safety endpoints: physical exam | Day 0 to day 84
  Abnormal physical examination
Safety endpoints: ECG | Day 0 to day 84
  Abnormal Electrocardiogram (ECG)
Safety endpoints: labs | Day 0 to day 84
  Number of abnormal results of Hematology, Biochemistry and Urinalysis

SECONDARY OUTCOMES:
Incidence rate of Acute kidney injury | from baseline up to 72 hours after PCI procedure
  definition of CI-AKI: Serum Creatinine absolute variation ≥ 0.5mg/dL or Serum creatinine relative variation increasing 25% from baseline up to 72 hours after CAG with the exposure of contrast medium and PCI
Long term kidney function: Serum creatinine | week 4 and week 12
  Serum creatinine level
Long term kidney function: eGFR | week 4 and week 12
  eGFR level
Kidney function parameters: creatinine, BUN | over 12-week period
  Serum creatinine and BUN level
Kidney function parameters: eGFR | over 12-week period
  eGFR using CKD-EPI
pharmacokinetics parameters: the area under the plasma concentration-time curve (AUC0-last, AUCtau) | Day -2~2
  to be assessed from plasma and urine samples (subset of subjects only)
pharmacokinetics parameters: peak concentration (Cmax, Tmax) | Day -2~2
  to be assessed from plasma and urine samples (subset of subjects only)
pharmacokinetics parameters: steady state peak plasma concentration (Css,max) | Day -2~2
  to be assessed from plasma and urine samples (subset of subjects only)
pharmacokinetics parameters: steady state trough plasma concentration (Css,min) | Day -2~2
  to be assessed from plasma and urine samples (subset of subjects only)
pharmacokinetics parameters: steady state after 5 consecutive days of drug administration | Day -2~2
  to be assessed from plasma and urine samples (subset of subjects only)
pharmacokinetics parameters: apparent total clearance (CL/F) | Day -2~2
  to be assessed from plasma and urine samples (subset of subjects only)
pharmacokinetics parameters: renal clearance (CLR) | Day -2~2
  to be assessed from plasma and urine samples (subset of subjects only)
pharmacokinetics parameters: apparent nonrenal clearance (CLNR/F) | Day -2~2
  to be assessed from plasma and urine samples (subset of subjects only)
pharmacokinetics parameters: apparent volume of distribution (V/F) | Day -2~2
  to be assessed from plasma and urine samples (subset of subjects only)
pharmacokinetics parameters: terminal half-life (t1/2) | Day -2~2
  to be assessed from plasma and urine samples (subset of subjects only)
pharmacokinetics parameters: fraction/cumulated fraction of excreted in urine | Day -2~2
  to be assessed from plasma and urine samples (subset of subjects only)

OTHER OUTCOMES:
Biomarkers assessment | 72 hours
  NGAL, KIM-1, Cystatin-C and NT-proBNP
Composite PCI outcome | over 12-week period
  death, myocardial infarction (MI) and stent thrombosis (ST)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (2):
  - Florida Cardiovascular Research, Hialeah, Florida
  - Sarkis Clinical Trials, Ocala, Florida
- South Korea (12):
  - Kangwon National University Hospital, Chuncheon
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Inje University Ilsan Paik Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan